CLINICAL TRIAL: NCT07008534
Title: Evaluation of Neurosensory Function of Inferior Alveolar Nerve Following Lateralization With Sticky Bone Versus Nil Using Computer Guided Dental Implant Placement: A Randomized Clinical Trial
Brief Title: Inferior Alveolar Nerve Lateralization With Simultaneous Implant Placement in Atrophic Posterior Mandible
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Muhammad Ashraf Elsawi, Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IAN Lateralization
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Dental Implant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer guided immediate implant placement & IAN lateralization (Active Comparator): Patients receiving computer-guided immediate implant placement and inferior alveolar nerve (IAN) lateralization only.
  Interventions: Procedure: Patients receiving computer-guided immediate implant placement and inferior alveolar nerve (IAN) lateralization only.
- computer guided immediate implant placement & IAN lateralization with Sticky bone (Experimental): Patients receiving computer-guided immediate implant placement and inferior alveolar nerve (IAN) lateralization with sticky bone
  Interventions: Procedure: IAN lateralization with computer-guided immediate implant placement using Sticky Bone

INTERVENTIONS:
Procedure: Patients receiving computer-guided immediate implant placement and inferior alveolar nerve (IAN) lateralization only. — Standard procedure without Sticky Bone application.
  Arms: Computer guided immediate implant placement & IAN lateralization
Procedure: IAN lateralization with computer-guided immediate implant placement using Sticky Bone — The same as the control with additional application of Sticky Bone as an insulator for enhanced neurosensory disfunction
  Arms: computer guided immediate implant placement & IAN lateralization with Sticky bone

SUMMARY:
The aim of this study is to evaluate the effect of sticky bone on acceleration of recovery of the neurosensory dysfunction of the inferior alveolar nerve following inferior alveolar nerve lateralization surgery for implant placement in patients with posterior vertical bone deficiency in order to overcome the main disadvantage of this technique & provide a reliable,saving time - computer guided simultaneous implant placement- and improved technique.

DETAILED DESCRIPTION:
Lateralization of IAN allows simultaneous implant placement with longer implants and primary stability.2 IAN lateralization provides an option to avoid costly, prolonged bone graftt and also healing periods can be reduced by this option of treatment Vestibular depth remains intact as there is no augmentation in the underlying bone defect. 2 IAN lateralization technique has also some advantages such as less morbidity and less of peri-implant disease.2 In case of the IAN is located in the superior part of the body of the mandible , and presence of mild atrophy of the edentulous alveolar ridge will fetch the alveolar ridge in a close relation to the neuro-vascular bundle, The incidence of "high" IAN locations ranges from 14.6 to 30.7%. 1However there is some complications such as numbness after surgery which is considered as the most common one also prevent thermal conductivity via implants(Kahnberg et al., 2000) so sticky bone is going to be used to act as an insulator between dental imlants & Inferior alveolar nerve and it contains a number of growth factors so it is predicted to play an important role to enhance recovery of the inferior alveolar nerve after surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring oral rehabilitation with dental implants in vertically atrophied

  * Posterior mandibular region, less than 8mm of bone above the mandibular canal.
  * Patients should be free from any systemic conditions that may affect normal healing.
  * Absence of any pathological conditions involving mandibular bones.

Exclusion Criteria:

* Patients under bisphosphonates treatment.

  * Any contraindication for general anaesthesia.
  * Osteoporotic patients.
  * Patients with neurological disorders (neuralgias, Parkinson' s disease).
  * Patients with systematic disease that may complicate healing.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical neurosensory assessment of inferior alveolar nerve. | 6 months

IPD SHARING:
Plan to Share IPD: Undecided